CLINICAL TRIAL: NCT06450535
Title: Radiographic and Histological Assessment of Retromolar Autogenous Onlay Bone Block Versus Cortical Shell for Augmentation of Horizontally Deficient Anterior Maxilla: (Randomized Clinical Trial).
Brief Title: Radiographic and Histological Assessment of Autogenous Onlay Block Versus Cortical Shell on Anterior Maxilla
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maria Ibrahim Nageeb, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD_CU_2024_26_1
Record Dates: First submitted 2024-05-09; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Alveolar Bone Loss
Keywords: Autogenous onlay bone block; Cortical shell technique
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Randomzed cinical trial
  A trial will be caried out in hosptal of Oral and Maxllolacial surgery department- Faculy of Oral and Dental Medicine Cairo Univerity.
  Equal randomizaion: participants wih equal probabilites for intervenion
  Postive controlled :Both groups receiving treatment
  Parallel group study: Each group of patients receives a single treatment simutaneously
Who Masked: Participant
Masking Description: This trial is considered a randomized single blind clinical trial due to the following:
  * The participants will be blinded to the technique that will be used during the surgical procedure.
  * The operator will not be blinded for both techniques during the surgical procedure as the two techniques are different.
  * The outcome assessor cannot be blinded. C) Data collection, management, and analysis:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous onlay block from retromolar bone (Experimental): In the first intervention, a bone block harvested from the donor site was fixed with osteosynthesis titanium screws to the recipient site as an onlay graft to achieve a horizontal enlargement of the alveolar ridge.
  ● Placement of the bone graft was always guided by an augmentation template
  Interventions: Procedure: Autogenous onlay bone block harvesting from retromolar bone in anterior maxilla
- Cortical shell technique from retromolar bone (Active Comparator): The harvested cortical plate was then split longitudinally in two parts using a microsaw, and thinned with the bone scraper to achieve a plate of 1 mm thickness.
  * The plate was fixed at a distance from the residual ridge with 2 screws.
  * Autogenous bone particles, collected with the bone scraper, were tightly packed into the gap between the plate and the recipient site.
  Interventions: Procedure: Autogenous cortical shell technique from retromolar bone in anterior maxilla

INTERVENTIONS:
Procedure: Autogenous onlay bone block harvesting from retromolar bone in anterior maxilla — Surgical protocol ( retromolar bone harvesting) After injecting local anesthesia a crestal incision is done, from a point on the occlusal surface along the external oblique ridge and extending anteriorly and inferiorly through the buccal mucosa, parallel to the gingival margin of the mandibular molars.
  The subperiosteal dissection extend to expose the ascending ramus and the retromolar region With the aid of surgical carbide burs, two proximal vertical cuts penetrating the cortex of the external oblique ridge.
  The depth of penetration of the posterior cut did not exceed 2.5 mm to avoid injury to the inferior alveolar nerve.
  By using microsaw , an inferior cut of 3.2 mm in depth joining the anterior and posterior vertical cuts was done.
  Small perforations of 3-4 mm in depth were performed on the superior aspect of the external oblique ridge using 1 mm drill bur.
  Finally, the block was sheared off using a chisel.
  Other Names: Autogenous onlay block from retomolar bone
  Arms: Autogenous onlay block from retromolar bone
Procedure: Autogenous cortical shell technique from retromolar bone in anterior maxilla — The harvested cortical plate was then split longitudinally in two parts using a microsaw, and thinned with the bone scraper to achieve a plate of 1 mm thickness.
  The plate was fixed at a distance from the residual ridge with 2 screws. Autogenous bone particles, collected with the bone scraper, were tightly packed into the gap between the plate and the recipient site.
  Other Names: Cortical shell technique from retromolar bone
  Arms: Cortical shell technique from retromolar bone

SUMMARY:
Two groups of patient with horizontally deficient anterior maxilla indicated for bone augmentation ,one will be subjected to autogenous onlay bone block from retromolar bone and the other to cortical shell from retromolar bone also.

DETAILED DESCRIPTION:
* Two groups of patients with horizontally deficient anterior maxilla indicated for bone augmentation, the first group will be subjected to autogenous onlay bone block from retromolar bone and the other group to cortical shell from retromolar bone also.
* periodontal therapy will be performed before any procedure and oral hygiene measures will be given to the patient.
* After injecting local anesthesia in the anterior maxillary region a trapezoidal flap will be performed in the area of horizontal bone defect (the recipient site).
* The recipient site will be decorticated and recontoured using a round bone bur for better adaptation of the graft and to improve graft-to-recipient bone contact.
* Bone harvesting will be carried out from retromolar region (the donor site) a crestal incision will be carried out 5 mm below and parallel to the gingival margin of the mandibular molars.
* subperiosteal dissection will be extended to expose the ascending ramus and the retromolar region.
* Using piezoelectric device a crestal cut and two proximal vertical cuts penetrating the cortex of the external oblique ridge will be performed then the inferior cut will be carried out.
* Using a mallet and chisel the bone block will be sheared off.
* The underlying cancellous bone will be gently retrieved and the collected bone will be conserved in sterile saline, followed by suturing the mucosal wound.
* Onlay bone block graft procedure (control group)
* In the first intervention, a bone block harvested from the donor site will be fixed with osteosynthesis titanium screws to the recipient site as an onlay graft to achieve a horizontal enlargement of the alveolar ridge.
* Cortical shell graft procedure (intervention group)
* The harvested cortical plate will be split longitudinally in two parts using a micro-saw and thinned with the bone scraper to achieve a plate of 1 mm thickness.
* The plate will be fixed at a distance from the residual ridge with 2 screws.
* Autogenous bone particles, collected with the bone scraper, were tightly packed into the gap between the plate and the recipient site.
* Radiographic assessment will be achieved by CBCT scan immediately and 4 months postoperatively to evaluate bone regeneration and final horizontal bone width.
* In the two groups, the screws will be removed 4 months postoperatively after final CBCT.
* The bone formed in the gap between the bone segment and the original bone will be measured from the CBCT scan.
* Before the intraoperative installment of the dental implants, bone core biopsies will be retrieved from each patient's recipient sites followed by implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients in both sex with partial edentulism of the maxilla and requiring horizontal ridge augmentation
* The ages of the patients ranged from 20 to 60 years.
* The residual ridge width in these patients are less than 4.m
* Sufficient bone in intra-oral donor sites are available (external oblique ridge)
* Patients free from any systemic conditions and bone metabolism diseases that might interfere with the surgical intervention, soft tissue or hard tissue healing.
* The vertical level should be in a favourable esthetic appearance with normal inter-arch space
* The minimum number of missing teeth in the anterior maxilla alveolar ridge is one single extracted teeth

Exclusion Criteria:

* Subjected to irradiation in the head and neck area less than 1 year before implantation.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
radiographic analysis | 4 month postoperative
  calculation of bone width gain using cone beam computed tomography

SECONDARY OUTCOMES:
histomorphometric analysis | 4 months postoperative
  to assess the bone quality for each technique

CONTACTS AND LOCATIONS:
Overall Officials: mohamed atef, PhD, Study Director — faculty of oral and dental medicine,cairo university
Locations (1):
- faculty of oral and dental medicine ,Cairo university, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Breakage of internal maxillary distractor: considerable complication of maxillary distraction osteogenesis — http://pubmed.ncbi.nlm.nih.gov/18585604/
- See also: The outcome of intraoral onlay block bone grafts on alveolar ridge augmentations: A systematic review — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4393991/
- See also: Lateral Ridge Augmentation Using Autogenous Block Grafts and Guided Bone Regeneration: A 10-Year Prospective Case Series Study — http://pubmed.ncbi.nlm.nih.gov/27476677/
- See also: Vertical Distraction Osteogenesis of Edentulous Ridges for Improvement of Oral Implant Positioning: A Clinical Report of Preliminary Results. — http://www.researchgate.net/publication/12053873_Vertical_Distraction_Osteogenesis_of_Edentulous_Ridges_for_Improvement_of_Oral_Implant_Positioning_A_Clinical_Report_of_Preliminary_Results
- See also: Long-Term Results of Peri-implant Conditions in Periodontally Compromised Patients Following Lateral Bone Augmentation. — http://pubmed.ncbi.nlm.nih.gov/28095518/
- See also: Augmentation of the sinus floor with mandibular bone block and simultaneous implantation: a 6-year clinical investigation — http://pubmed.ncbi.nlm.nih.gov/10453672/
- See also: "Secure and effective stabilization of different sized autogenous bone grafts." — http://www.stoma.de/fileadmin/user_upload/Downloads/Fachbeitraege/JOS_microscrew_Khoury_Hidajat.pdf
- See also: Mechanisms of guided bone regeneration: a review — http://pubmed.ncbi.nlm.nih.gov/24894890/
- See also: Evolution of Barrier Membranes in Periodontal Regeneration-"Are the third Generation Membranes really here? — http://pubmed.ncbi.nlm.nih.gov/25654055/
- See also: Treatment concepts of horizontally deficient ridges-A retrospective study comparing narrow-diameter implants in pristine bone with standard-diameter implants in augmented bone. — http://pubmed.ncbi.nlm.nih.gov/34224171/
- See also: Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. — http://pubmed.ncbi.nlm.nih.gov/12956475/
- See also: The edentulous ridge expansion technique: a five-year study. — http://pubmed.ncbi.nlm.nih.gov/7751111/